CLINICAL TRIAL: NCT03452943
Title: A Randomized, Double-blind, Placebo-controlled Study of TEV-50717 (Deutetrabenazine) for the Treatment of Tourette Syndrome in Children and Adolescents
Brief Title: Alternatives for Reducing Tics in Tourette Syndrome (TS): A Study of TEV-50717 (Deutetrabenazine) for the Treatment of Tourette Syndrome in Children and Adolescents
Acronym: ARTISTS1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Nuvelution TS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV50717-CNS-30046; 2016-000622-19 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; adolescents; children
MeSH Terms: conditions — Tourette Syndrome | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEV-50717 (Experimental): TEV-50717 tablets twice daily (BID) up to 48 milligrams (mg)/day orally for a total of 12 weeks
  Interventions: Drug: TEV-50717; Drug: Placebo
- Placebo (Placebo Comparator): Placebo matched to TEV-50717 BID for a total of 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-50717 — 6, 9, 12, 15, and 18 mg oral tablets
  Other Names: Deutetrabenazine
  Arms: TEV-50717
Drug: Placebo — Placebo matched to TEV-50717 tablets will be taken BID for 12 weeks.

SUMMARY:
This is a study to evaluate the efficacy and safety of deutetrabenazine (TEV-50717) tablets for the reduction of motor and phonic tics associated with TS in children and adolescents 6 through 16 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 6 to 16 years of age, inclusive.
* Participant weighs at least 44 pounds (20 kilograms [kg]).
* The participant's active tics are causing distress or impairment.
* Participant is able to swallow study medication whole.
* Participant is in good general health.
* Women/girls of childbearing potential whose male partners are of childbearing potential must use contraception for the duration of the study.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participant has a neurologic disorder other than TS that could obscure the evaluation of tics.
* Participant has a confirmed diagnosis of bipolar disorder, schizophrenia, or another psychotic disorder.
* Participant has clinically significant depression at screening or baseline.
* Participant has a history of suicidal intent or related behaviors within 2 years of screening.
* Participant has a history of a previous actual, interrupted, or aborted suicide attempt.
* Participant has a first-degree relative who has completed suicide.
* Participant has received comprehensive behavioral intervention for tics (CBIT) for TS or cognitive behavioral therapy (CBT) for obsessive-compulsive disorder (OCD) within 4 weeks of screening.
* Participant has an unstable or serious medical illness at screening or baseline.
* Participant is pregnant or breastfeeding.

  * Additional criteria apply, please contact the investigator for more information.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (42):
- United States (27):
  - Teva Investigational Site 046-0104, Dothan, Alabama
  - Teva Investigational Site 046-0117, Sun City, Arizona
  - Teva Investigational Site 046-0107, Rogers, Arkansas
  - Teva Investigational Site 046-0126, Anaheim, California
  - Teva Investigational Site 046-0101, Sacramento, California
  - Teva Investigational Site 046-0111, San Diego, California
  - Teva Investigational Site 046-0130, Santa Ana, California
  - Teva Investigational Site 046-0132, Miami, Florida
  - Teva Investigational Site 046-0115, Orlando, Florida
  - Teva Investigational Site 046-0114, St. Petersburg, Florida
  - Teva Investigational Site 046-0116, Atlanta, Georgia
  - Teva Investigational Site 046-0133, Naperville, Illinois
  - Teva Investigational Site 046-0128, Boston, Massachusetts
  - Teva Investigational Site 046-0110, Saint Charles, Missouri
  - Teva Investigational Site 046-0134, Lincoln, Nebraska
  - Teva Investigational Site 046-0109, Voorhees Township, New Jersey
  - Teva Investigational Site 046-0124, New York, New York
  - Teva Investigational Site 046-0102, Rochester, New York
  - Teva Investigational Site 046-0112, Rochester, New York
  - Teva Investigational Site 046-0125, Raleigh, North Carolina
  - Teva Investigational Site 046-0106, Oklahoma City, Oklahoma
  - Teva Investigational Site 046-0113, Dallas, Texas
  - Teva Investigational Site 046-0108, Houston, Texas
  - Teva Investigational Site 046-0103, Houston, Texas
  - Teva Investigational Site 046-0120, San Antonio, Texas
  - Teva Investigational Site 046-0105, Orem, Utah
  - Teva Investigational Site 046-0118, Petersburg, Virginia
- Canada (2):
  - Teva Investigational Site 046-0201, Ajax, Ontario
  - Teva Investigational Site 046-0202, Ottawa, Ontario
- Denmark (2):
  - Teva Investigational Site 046-0302, Herlev
  - Teva Investigational Site 046-0301, Odense
- Russia (3):
  - Teva Investigational Site 046-0702, Stavropol
  - Teva Investigational Site 046-0704, Tomsk
  - Teva Investigational Site 046-0703, Voronezh
- Serbia (3):
  - Teva Investigational Site 046-1702, Belgrade
  - Teva Investigational Site 046-1703, Belgrade
  - Teva Investigational Site 046-1701, Novi Sad
- Spain (5):
  - Teva Investigational Site 046-0604, Barcelona
  - Teva Investigational Site 046-0605, Madrid
  - Teva Investigational Site 046-0602, Madrid
  - Teva Investigational Site 046-0603, Málaga
  - Teva Investigational Site 046-0601, Seville

REFERENCES:
- [Derived] Jankovic J, Coffey B, Claassen DO, Jimenez-Shahed J, Gertz BJ, Garofalo EA, Stamler DA, Wieman M, Savola JM, Gordon MF, Alexander J, Barkay H, Harary E. Safety and Efficacy of Flexible-Dose Deutetrabenazine in Children and Adolescents With Tourette Syndrome: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2128204. doi: 10.1001/jamanetworkopen.2021.28204. PMID 34609495

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 119 participants were randomized in a 1:1 ratio to either TEV-50717 or placebo group.
Groups:
- TEV-50717: Participants received TEV-50717 as oral tablets at a starting dose of 6 milligrams (mg)/day, with the dose titrated weekly for 7 weeks to an optimal level. The target maximum daily dose was determined by body weight and cytochrome P450 2D6 (CYP2D6) impairment status at baseline. Maximum total daily dose for participants greater than or equal to (≥) 40 kilograms (kg) was 48 mg/day (24 mg twice daily [BID]), 30 to less than (<) 40 kg was 42 mg/day (21 mg BID), and 20 to <30 kg was 30 mg/day (15 mg BID). For those considered CYP2D6 impaired, maximum daily dose for participants ≥40 kg was 36 mg/day, 30 to <40 kg was 24 mg/day, and 20 to <30 kg was 18 mg/day. Total daily doses of ≥12 mg/day was divided into a BID administration. Depending on the dose, TEV-50717 tablets and/or placebo tablets were taken to maintain the blind. Participants then received TEV-50717 at the optimal level as maintenance therapy daily for 5 weeks.
- Placebo: Participants received placebo matched to TEV-50717 BID for a total of 12 weeks.
Period: Titration Period (7 Weeks)
Arm/Group | TEV-50717 | Placebo
Started (Intent-to-treat (ITT) analysis set: all randomized participants) | 59 | 60
Safety Analysis Set (Received at least 1 dose of study drug) | 58 | 59
Modified ITT (mITT) Analysis Set (Received at least 1 dose of study drug; had both baseline & at least 1 postbaseline YGTSS assessment) | 58 | 59
Completed | 54 | 56
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Period: Maintenance Period (5 Weeks)
Arm/Group | TEV-50717 | Placebo
Started | 54 | 56
Completed | 51 | 56
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants.
Groups:
- TEV-50717: Participants received TEV-50717 as oral tablets at a starting dose of 6 mg/day, with the dose titrated weekly for 7 weeks to an optimal level. The target maximum daily dose was determined by body weight and CYP2D6 impairment status at baseline. Maximum total daily dose for participants ≥40 kg was 48 mg/day (24 mg BID), 30 to <40 kg was 42 mg/day (21 mg BID), and 20 to <30 kg was 30 mg/day (15 mg BID). For those considered CYP2D6 impaired, maximum daily dose for participants ≥40 kg was 36 mg/day, 30 to <40 kg was 24 mg/day, and 20 to <30 kg was 18 mg/day. Total daily doses of ≥12 mg/day was divided into a BID administration. Depending on the dose, TEV-50717 tablets and/or placebo tablets were taken to maintain the blind. Participants then received TEV-50717 at the optimal level as maintenance therapy daily for 5 weeks.
- Total: Total of all reporting groups
Arm/Group | TEV-50717 | Placebo | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (2.52) | 11.5 (2.59) | 11.5 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 53 | 51 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 51 | 50 | 101
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 53 | 102
  Black | 3 | 3 | 6
  Asian | 1 | 1 | 2
  Native American | 1 | 0 | 1
  Multiple | 3 | 1 | 4
  Other | 2 | 2 | 4
Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) [Mean (Standard Deviation); unit: units on a scale] — YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 for severe). Motor tic severity score (MTSS) is the sum of 5 items for motor tic severity and vocal tic severity score (VTSS) is the sum of 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome.
  units on a scale | 31.7 (5.81) | 33.0 (5.96) | 32.3 (5.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the TTS of the YGTSS at Week 12
Description: YGTSS rating scale is a semi-structured clinician rating instrument that provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic tics. YGTSS is composed of 11 items: 5 items for motor tic severity, 5 items for vocal tic severity, and 1 item for impairment. Each item for motor tic severity and vocal is rated on a 6-point scale (0 for none to 5 to severe). MTSS is the sum of the 5 items for motor tic severity and VTSS is the sum of the 5 items for vocal tic severity. TTS is the sum of MTSS and VTSS, ranges from 0 (none/absent) to 50 (severe). Higher scores indicate greater severity/worse outcome. Least square (LS) mean and standard error (SE) was calculated using mixed-model repeated-measures (MMRM) with treatment group, week (5 levels: weeks 2, 4, 6, 9, and 12), and the treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6 to 11 years, 12 to 16 years) as covariates.
Time Frame: Baseline, Week 12
Population: mITT analysis set included all randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline YGTSS assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale | -9.1 (1.28) | -8.4 (1.25)
Statistical Analysis 1: Comparison: TEV-50717 vs Placebo; Test type: Other; p = 0.692, Mixed Models Analysis — Threshold for significance at 0.05 level; LS mean difference = -0.7, 95% CI 2-sided [-4.1 to 2.8]

2. Secondary Outcome: Change From Baseline in the Tourette Syndrome-Clinical Global Impression (TS-CGI) Score at Week 12
Description: The TS-CGI scale is a 7-point Likert scale that allows the clinician to use all available information to assess the impact of tics on the participant's quality of life. The TS-CGI is rated as follows: 1 (normal or no tics at all), 2 (borderline), 3 (mild), 4 (moderate), 5 (marked), 6 (severe), and 7 (extreme, incapacitating tics). Lower scores indicate better quality of life. LS mean and SE was calculated using MMRM with treatment group, week (5 levels: weeks 2, 4, 6, 9, and 12), and the treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6 to 11 years, 12 to 16 years) as covariates.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale | -0.7 (0.13) | -0.7 (0.12)

3. Secondary Outcome: Change From Baseline in the Tourette Syndrome-Patient Global Impression of Impact (TS-PGII) Score at Week 12
Description: The TS-PGII is a single-item questionnaire that asks the participant to assess the degree of impact due to current tics (How much do your current tics disrupt things in your life?). The TS-PGII uses a 5-point scale, ranging from not at all (1) to very much (5), to assess overall response to therapy.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale | -0.7 (0.18) | -0.4 (0.14)

4. Secondary Outcome: Change From Baseline in the Child and Adolescent Gilles de la Tourette Syndrome - Quality of Life (C&A-GTS-QOL) Activities of Daily Living (ADL) Subscale Score at Week 12
Description: C&A-GTS-QOL is a 27-item questionnaire that asks participant to assess the extent to which their quality of life is impacted by their symptoms. C&A-GTS-QOL contains 6 subscales (cognitive, coprophenomena, psychological, physical, obsessive-compulsive, and ADL) and uses a 5-point Likert scale ranging from no problem to extreme problem. Following 3 questions from 27-item questionnaire were assessed in ADL C&A-GTS-QOL subscale: Question 2 (Had difficulty with school or sport activities?), 24 (Felt you needed more help or support from other people?), and 26 (Had difficulty going out with other people?). Total score of ADL subscale ranged from 0 (no problem) to 12 (extreme problem). Lower score indicated better quality of life. LS mean and SE was calculated using MMRM with treatment group, week (5 levels: weeks 2, 4, 6, 9, and 12), and treatment group by week interaction as fixed effects; and baseline TTS, region, and age group at baseline (2 levels: 6-11 years, 12-16 years) as covariates.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEV-50717 | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale | -9.9 (2.37) | -8.8 (2.27)

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) to follow-up (Week 14)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TEV-50717 | Placebo
Number analyzed (Participants) | 58 | 59
percentage of participants
  Any AEs | 65.5 | 55.9
  Treatment-related AEs | 50.0 | 20.3
  Serious AEs | 0 | 0
  AEs leading to discontinuation | 1.7 | 1.7

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to follow-up (Week 14)
Description: Safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | TEV-50717 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 22/58 | 23/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEV-50717 (N=58) | Placebo (N=59)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (11)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Fatigue (General disorders) | 7 (8) | 3 (4)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 7 (9)
Weight increased (Investigations) | 7 (7) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 6 (12)
Somnolence (Nervous system disorders) | 5 (8) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Depressed mood (Psychiatric disorders) | 2 (2) | 3 (3)
Enuresis (Psychiatric disorders) | 4 (6) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT03452943/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03452943/SAP_001.pdf